CLINICAL TRIAL: NCT02477241
Title: Study of Brain Areas Involved in the Sensation of Bladder Filling in Healthy Females and Untreated Females With Overactive Bladder (OAB) Using fMRI and Water Pressure Urodynamics
Brief Title: Brain Areas Involved in Bladder Filling and Contraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Sajjad Rahmana'i, M.D. PhD, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL52605.068.15
Record Dates: First submitted 2015-05-20; First posted 2015-06-22 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Urinary Bladder, Overactive
Keywords: overactive bladder syndrome; urgency urinary incontinence; fMRI; urodynamics
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy female subjects (Other): Healthy female subjects with or without overactive bladder undergoing functional MRI brain and urodynamic study.
  Interventions: Procedure: Uroflowmetry; Device: fMRI

INTERVENTIONS:
Procedure: Uroflowmetry — A cystometric test measures how much urine the bladder can hold, how much pressure builds up inside the bladder as it stores urine, and how full it is when the urge to urinate begins. Uroflowmetry is the measurement of urine speed and volume.
  Other Names: urodynamic investigation
Device: fMRI — Functional magnetic resonance imaging or functional MRI (fMRI) is a functional neuroimaging procedure using MRI technology that measures brain activity by detecting associated changes in blood flow. This technique relies on the fact that cerebral blood flow and neuronal activation are coupled. When an area of the brain is in use, blood flow to that region also increases.

SUMMARY:
Overactive Bladder syndrome (OAB) is a medical condition with symptoms of urgency, with or without incontinence, usually with frequency and nocturia, with no proven infection or obvious pathology 1. This study will explore the relationship between OAB, obstruction and the micro contractions as well as the brain areas involved in both normal desire to void and urgency, gaining a better understanding of the bladder pathophysiology and in the future allowing better strategy of treatment options for patients suffering from OAB.

DETAILED DESCRIPTION:
Overactive Bladder Syndrome The International Continence Society (ICS) has defined Overactive Bladder syndrome (OAB) as a medical condition with symptoms of urgency, with or without incontinence, usually with frequency and nocturia, with no proven infection of obvious pathology.

OAB has an overall prevalence in Western Europe and the United States of 16% to 17%. Epidemiological evidence indicates that symptoms of OAB are common and likely to affect up to 50-100 million persons worldwide. In the EPIC study which was conducted in 5 countries in > 19000 men and women aged > 18 years, using the ICS definitions for OAB, the prevalence of OAB was 10.8% in men and 12.8% in women, and its prevalence increased with age. The prevalence in women for storage was 59.2%, in voiding 19.5% and in post micturition symptoms 14.2%.

The fundamental symptom is urgency, which is widely considered to be the driver of other urological symptoms. Urgency is a sudden compelling desire to pass urine, which is difficult to defer. The urological symptoms can have a considerable negative impact on quality of life, typically resulting in embarrassment and loss of dignity, which might affect relationships, intimacy and self-image.

Conventional urodynamic test Diagnostic testing of lower urinary tract function by performing urodynamic investigations is currently widely accepted. The aim of the clinical urodynamics is to produce symptoms whilst making precise measurements in order to identify underlying causes for the symptoms and to quantify the related pathophysiological processes. Urodynamics allows direct assessment of lower urinary tract function by the measurement of physiological parameters (e.g. voiding pressure parameters; minimal urethral opening detrusor pressure and urethral resistance factor), micturitions volume and leakage volume).

Urodynamics cannot be performed as an automated protocol due to current limitations of urodynamic equipment and the lack of consensus on the precise method of measurement, signal processing, quantification, documentation and interpretation. The Good Urodynamic Practices developed by ICS provides guidelines regarding the strategy for urodynamic measurement, equipment set up and configuration, signal testing, plausibility controls, pattern recognition, and artefact correction.

During cystometry, involuntary detrusor contractions can only be found in 40% to 60% of patients with OAB symptoms. Detrusor overactivity contractions can occur either during filling or at the end. Conventional urodynamic remains the gold standard for investigating lower urinary tract dysfunction.

Functional Magnetic Resonance Imaging fMRI is an imaging modality that has recently been further developed to study the different parts of the human body through blood flow changes. In close collaboration with Maastricht University, Scannexus has made multiple 7 Tesla MRI scans available for our study in order to gain further insight into brain functioning areas.

Bladder Sensations Most of the understanding on the experience of bladder sensation during filling in normal individuals is based upon the work of Wyndaele and De Wachter. The sensation scoring system developed seek to determine the underlying reasons an individual patient usually void and is not meant to serve as an index of urgency or severity. The 4-point scoring scale ranges from voiding out of convenience (no urgency=0) to desperate urgency score=3) to capture perception of urgency on a continuum rather per se. The condition is recognised clinically as the 'Overactive Bladder (OAB) Symptom Complex'. It is associated with increased sensations to void which result in an increased voiding frequency, as determined from voiding diaries. OAB is further characterised during cystometric investigation by the occurrence of involuntary contractions of the bladder during the filling phase and, typically in the 'full bladder' by a strong sensation described as 'urgency' (a strong compelling desire to void that cannot be deferred which is more intense than a normal urge to void).

Overactive bladder syndrome (OAB) is associated with episodic increased bladder sensations to void, which result in increased in voiding frequency. During cystometric investigations, OAB is also characterised by the occurrence of involuntary bladder contractions during the filling phase and typically in the full bladder, a strong sensation described as urgency (described as a strong compelling desire to void that cannot be deferred and is more intense than the normal urge to void). It is during these urgency episodes that leakages (urgency incontinence) sometimes occur. In 46% of patients with the sensation of urgency, it is associated with bladder contractions.

Many studies investigated the link between patient reported sensations and bladder properties using standard rapid fill cystometry. This leads to the concept that bladder sensation is episodic. These episodic sensations are supposedly greater in patients with OAB and occur in lower bladder volumes, thus generating the sensation of urgency and more frequent voiding.

As described in literature sensations associated with bladder filling were different from those of imminent voiding. The sensations during filling were associated with a generalised feeling in the lower abdomen while the more intense sensations of imminent pre-void were located deeper down in the urethra. This anatomical variation may reflect different sensations and different underlying mechanisms. This supports that there are two systems generating sensation: 'continuous sensation' associated with the early filling phase and intense phasic sensations associated with the urethra.

An alternative view of bladder sensation was formulated many years ago. It proposes that the information from the bladder is generated continuously and that an awareness of bladder volumes is available through the entire filling phase. This is supported by neuro-physiological data demonstrating an almost continuous afferent outflow from the bladder receptors as the bladder fills. As a conclusion the physiological bases of the sensation or "urge" or "urgency" is still unknown.

Moreover, patients with OAB with or without detrusor overactivity (DO) on urodynamics all have in common that they have a sense of urgency. This sense is described as a sudden, compelling desire to void, which cannot be postponed. Affected individuals have the fear to loose urine (incontinence) and some even actually do. It is still not known if the same brain areas are involved in a normal desire to void in controls, as in OAB patients both with and without DO when they feel urgency. In our study we would like to answer this question by conducting simple urodynamics during an fMRI scan while the patient's bladder is filled through normal diuresis and their sense of urgency is registered through a push button.

In the past a few studies have been conducted with the fMRI of the central nervouse system in relation to bladder control. Poor bladder control has been reported to be specifically associated with inadequate activation of orbitofrontal cortex. Clinically, frontal cortical lesions are known to cause bladder control problems.. In addition, urinary urgency in patients with OAB was shown to be associated with increased activation of the limbic cortex through fMRI studies in women with OAB. A more recent study with fMRI showed that there were significant and vast changes in the brain's functional connectivity when bladder is filled, suggesting that the central process responsible for the increased control during the full bladder state appears to largely rely on the how distributed brain systems. In all these studies, a 3 Tesla fMRI has been used. The 7 Tesla fMRI which is intended to be used in our study will enable us to study brain areas that are more difficult to assess with 1,5 and 3 Tesla.

Moreover, none of the previous studies have included a protocol to measure bladder pressure, bladder sensation and fMRI scans of the brain simultaneously.

ELIGIBILITY:
Healthy Subjects

Inclusion Criteria:

* Healthy female subjects above 18 years of age.
* Has provided written informed consent prior to any study related procedures.

Overactive bladder patients

Inclusion Criteria:

* Female subjects above 18 years of age.
* Has provided written informed consent prior to any study related procedures.
* History of signs and symptoms of OAB including urinary frequency, urgency or urge incontinence for greater than or equal to 3 months.
* At the screening visit, the subject should be either naïve to OAB treatment (e.g. no prior history of medications to treat lower urinary tract symptoms (LUTS), including OAB) or currently on treatment for LUTS (including OAB) and is willing to undergo a washout period for 3 weeks.

Healthy subjects:

Exclusion Criteria:

1. History of lower urinary tract symptoms (LUTS), including OAB.
2. History of stress urinary incontinence, urethral sphincter incompetence and neurogenic detrusor overactivity.
3. History of signs or symptoms suggestive of urinary tract infection (confirmed by positive urine analysis).
4. History of bladder outlet obstruction (not including detrusor-overactivity) for example bladder/vesico-uterine prolapse (> grade II) or chronic obstruction.
5. History of urinary tract surgery less than or equal to 6 months prior to screening.
6. Has an indwelling catheter or permanent catheter fitted.
7. History of pelvic area radiotherapy treatment.
8. Uncontrolled diabetes mellitus.
9. History of fibromyalgia.
10. Pregnant or intends to become pregnant during the study or sexually active, of childbearing potential and is unwilling to utilize a reliable method of birth control (note: reliable methods are contraceptive pills of combination type, hormonal implants, injectable contraceptives, sexual abstinence and vasectomized partner).
11. Pregnancy within 6 months before screening or breast feeding within 3 months before screening.
12. History of positive hepatitis A, B surface antigen, hepatitis C antibody or HIV test results.
13. Any use of drugs of abuse within 3 months prior to screening visit.
14. History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to screening visit.
15. History of drinking more than 14 units of alcohol per week within 3 months prior to screening visit.
16. Has any changes to prescribed medication or to dose of prescribed medication less than or equal to 1 month prior to screening which in the opinion of the Investigator, will interfere with the study procedures or compromise safety.
17. Is currently receiving or has a history of treatment with alpha blockers, beta receptor blockers or agonists, botulinum toxin (less than 12 months), resiniferatoxin or pelvic floor muscle relaxants less than or equal to 9 months prior to screening.
18. Any clinically significant abnormality following the investigator's review of screening physical examination.
19. Any clinically significant history of any other disease or disorder- gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the medical investigator.
20. Abnormal pulse and/or blood pressure measurements at the screening visit as follows: Pulse <40 or >90 bpm; systolic blood pressure >140 mmHg; diastolic blood pressure >90 mmHg; blood pressure and pulse measurements after subject has rested for 10 minutes.
21. Employees of the University of Maastricht involved in the study.
22. Claustrophobia, preventing a patient to have an fMRI scan
23. Patients with any metal implants in the body (except dental implants) that would prevent the patients to undergo fMRI scan.

For overactive bladder subjects Refer to healthy subjects exclusion criteria number 2 to number 23.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Bladder pressure changes during the filling phase with water pressure | up to two hours
  urodynamics during the fMRI study.

SECONDARY OUTCOMES:
HADS questionnaire (self-administered) screening for anxiety and depression | cross-sectional; filling out the HADS questionnaire (15 minutes)
  A secondary goal is to assess the correlation between bladder filling (Primary Outcome Measure) and subjects' bladder sensations in combination with psychological anxiety and depression status, which are both measured (screened for) through administering one questionnaire: the Hospital Anxiety and Depression Score (HADS) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gommert A. van Koeveringe, M.D. PhD, Principal Investigator — Maastricht University Medical Centre, Head of Department of Urology
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands